CLINICAL TRIAL: NCT07313553
Title: The Effect of Perineural Dexamethasone on Preventing Rebound Pain After Axillary Plexus Block in Hand Surgery
Brief Title: Prevention of Rebound Pain After Axillary Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, PROFESSOR, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMKO-CE-2023-004
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pain; Postoperative Care
Keywords: axillary nerve block; dexamethesone; rebound pain
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axillary Plexus Block with dexametasone (Active Comparator): In the cohort of patients undergoing hand surgery, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into intervention group. Intervention group will receive 30 ml of a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1%, containing 8 mg of dexamethasone.
  Interventions: Drug: Dexamathsone 4mg/ml associated with experimental arm
- Axillary Plexus Block control (Placebo Comparator): In the cohort of patients undergoing hand surgery, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into placebo group. Control group will receive a 30 ml of a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1%, containing 2 mL of saline solution.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Saline — 2 ml saline solution are added to 30 ml of a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1%
  Arms: Axillary Plexus Block control
Drug: Dexamathsone 4mg/ml associated with experimental arm — Intervention group will receive 30 ml of a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1%, containing 8 mg of dexamethasone.
  Arms: Axillary Plexus Block with dexametasone

SUMMARY:
This will be a single-center randomized double blind placebo control clinical trial. In the cohort of patients undergoing hand surgery under axillary nerve block, participants are recruited from those who are willing to consent and participate in the study, and will be randomly 1:1 divided into intervention group and placebo group.

DETAILED DESCRIPTION:
After the arrival to the operation room, monitoring including pulse oximetry, electrocardiogram, and noninvasive blood pressure was applied.

An 18 or 16-gauge IV cannula was inserted and Ringer's lactate infusion was started at a rate of 5 mL per kg per hour.

Antibioprophylaxis was systematically administered with 2 grams ofCefazolin 30 minutes before induction.

All patients were given an ultrasound-guided single-injection axillary plexus block by experienced anesthesiologists.

Sedation with 2 mg midazolam intravenously before block was administered.

In the group Dexamethasone (D), patients received axillary plexus block with a 30 ml of a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1%, containing 8 mg of dexamethasone.

In the group control (X), patients received a 30 mlof a 50/50 mixture of isobaric bupivacaine 0.5% and lidocaine 1% containing 2 ml saline solution.

For the axillary plexus block, patients were placed in a supine positionwith the arm in 90° of abduction and the forearm in flexion.A high frequency linear probe was placed on the transverse axis, over the axillary fold.The axillary artery, vein, and nerves surrounding the artery were visualized after scanning distally and proximally. The block needle (50 mm, 22G) was inserted in-plane from anterior to posterior, parallel to the ultrasound probe.It was advanced toward the musculocutaneous nerve (MCN) and local anesthetic was injected.Then, the needle was retracted and redirected deep relative to the axillary artery and local anesthetic was injectedaround the posterior aspect of the axillary artery and finallythe needle was retracted and redirected superficial to the axillary artery and local anesthetic was injected.

Before the surgical incision, the effectiveness of the sensory blockade of the axillary plexus was evaluated by a cold test in the different territories.

Post-operatively, all patients were put on systematic paracetamol 1 g every 6 hours, without exceeding 4 grams per day.

when the postoperative pain score (NRS) was >3/10, intravenous tramadol 100 mg was administered.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 75 years old.

  * Patients are current for hand surgery under axillary plexus block.
  * Patients classified ASA physical status I, II and III

Exclusion Criteria:

* - Contraindication to regional anesthesia.
* Patient's disapproval.
* Impaired cognition.
* Patients whose surgery must be done under general anesthesia (complex hand surgery or association of other)
* Allergy to paracetamol, dexamethasone or opioids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
incidence of Rebound pain | 1 hour postoperatively to 48 hours postoperatively
  The primary objective is the incidence of rebound pain, which was defined as severe pain (NRS ≥ 7) [Numerical rate scale from 0 no pain to 10 worst pain] at the surgical site during the first 48 hours postoperatively.

SECONDARY OUTCOMES:
Pain score at rest | hour 1, hour 48 postoperative
  Pain score at rest using NRS [Numerical Rate Scale from 0 no pain to 10 worst pain
Pain score at movement | hour 1, hour 48 postoperative
  Pain scores at mouvement using NRS [Numerical Rate Scale from 0 no pain to 10 worst pain
The analgesic consumption | hour 1, hour 24 postoperatively
  The number of rescue analgesic dose during the first 24 hours
Duration of motor block | hour 1 postoperatively, 12 hours after nerve block
  The end of motor block was defined by a total flexion of fingers and arm.
Blood glucose level | after nerve block, 24 hours after surgery
  level of glucose in serum blood